CLINICAL TRIAL: NCT05926037
Title: Evaluation of 3D Simulation and Planning of Left Atrial Appendage Occlusion Based on 3D Echocardiography
Acronym: USIM-LAAO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 23203_USIM-LAAO
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-06

CONDITIONS: ATRIAL APPENDAGE CLOSURE for ATRIAL FIBRILLATION

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare a semi-automatic 3D echocardiography-based left atrial appendix occlusion procedure planning with FEops, with other imaging modalities for evaluating the left atrial appendage dimensions and device prediction (sizing, deformation) pre-left atrial appendix occlusion , including the current "gold standard", CT- based FEops HEARTguideTM left atrial appendix occlusion procedure planning. A number of pre-specified endpoints are defined for analyzing this new approach.

DETAILED DESCRIPTION:
First, the investigator will compare dimensions of left atrial appendix ostium and device landing zone, and the predicted device size and deformation based on the gold standard (CT-based analysis by FEops HEARTguideTM, with ostium and landing zone dimensions, predicted device size (based on the device sizing chart) and device deformation predicted by FEops analysis of the 3D echo images. Complementary, dimensions and device size prediction derived from 3D echo-derived FEops analysis, will also be compared to measurements and device size prediction obtained from pre-procedural CT images and the 2D per-procedural transesophageal echocardiographic evaluation.

Secondly, the process of echo image analysis by FEops will be tested by evaluating the percentage of cases where FEops anatomical analysis is successful in providing a complete report. Based on the acquired 3D echo data, case processing is considered successful if ostium and landing zone diameters (minimum, maximum, mean and perimeter-based diameter), and device sizing, together with predicted device deformation, can be reported. The number of cases where only partial reporting is possible, as well the cases where no reporting is feasible, will also be recorded. If case analysis is not successful, the reason for failure will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for LAAO with an Amplatzer Amulet Left Atrial Appendage Occluder (Abbott Medical)
* clinical indication (in line with currently accepted indications and national reimbursement criteria)
* inclusion in 2 experienced Belgian LAAO centers (Brussels and Genk)

Exclusion Criteria:

* contra-indication for contrast (including contrast allergy and renal failure),
* contra-indication for radiation exposure (e.g. pregnancy)
* Inability by FEops to analyze CT images and provide a report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for LAAO with an Amplatzer Amulet Left Atrial Appendage Occluder (Abbott Medical) in 2 experienced Belgian LAAO centers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Level of agreement between dimensions (minimal, maximum, mean and perimeter-based diameter of ostium and landing zone) of FEops analysis based on 3D echocar-diography vs FEops analysis based on CT | DURING PROCEDURE

SECONDARY OUTCOMES:
Level of agreement between predicted device size by FEops analysis based on 3D echo vs FEops analysis based on CT | DURING PROCEDURE
Level of agreement between predicted device deformation by analysis based on 3D echo vs FEops analysis based on CT | DURING PROCEDURE
Level of agreement between dimensions (minimal, maximum, mean and perimeter-based diameter of ostium and landing zone) of FEops analysis based on 3D echo vs analysis based on 2D measurements on CT and peri-procedural echo | DURING PROCEDURE
Level of agreement between predicted device size by FEops analysis based on 3D echo vs FEops analysis based on 2D measurements on CT and peri-procedural echo | DURING PROCEDURE
The percentage of 3D echocardiography cases sent to FEops, where data on ostium and landing zone diameters, and device size prediction/deformation, can successfully be provided (descriptive) | DURING PROCEDURE
The percentage of 3D echocardiography cases sent to FEops, where data on ostium and landing zone diameters, and device size prediction/deformation, can only be par-tially, or are failed to be provided (descriptive) | DURING PROCEDURE
Most frequent reasons for failure to provide complete reporting after FEops analysis based on 3D echo images | DURING PROCEDURE

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Universitair Ziekenhuis Brussel, Jette

IPD SHARING:
Plan to Share IPD: No